CLINICAL TRIAL: NCT06772610
Title: The Efficacy and Safety of Ensartinib As Adjuvant Therapy in Stage I ALK-positive NSCLC Patients with High Risk Factors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chunxia Su, Director of Clinical Research Center, Shanghai Pulmonary Hospital, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024LY1286
Record Dates: First submitted 2025-01-10; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: NSCLC; ALK; Stage I; Adjuvant Treatment
Keywords: NSCLC; ALK positive; adjuvant treatment; high-risk factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Ensartinib 200 mg, once daily, orally, for a continuous period of 2 years.
  Interventions: Drug: Ensartinib group

INTERVENTIONS:
Drug: Ensartinib group — Ensartinib 200 mg, once daily, orally, for a continuous period of 2 years.

SUMMARY:
This study is designed to evaluate the efficacy and safety of a 2-year adjuvant treatment with Ensartinib in stage I ALK-positive non-small cell lung cancer (NSCLC) patients with high-risk factors. The study population includes patients with ALK-positive NSCLC who have undergone R0 resection and have not received any postoperative treatment, with a TNM stage of I and high-risk factors for recurrence.

DETAILED DESCRIPTION:
A total of 40 patients will be enrolled in the study. All patients will receive adjuvant therapy with Ensartinib at a dose of 200 mg, once daily, orally, for a continuous period of 2 years, or until disease recurrence or intolerable toxicity occurs. The efficacy and safety of Ensartinib treatment will be evaluated.Before any study-related procedures are conducted, informed consent will be obtained. Demographic information, a complete medical history, surgical history, and smoking history will be collected. The TNM stage of the primary tumor at diagnosis will be recorded/confirmed. Tumor assessments and other screening examinations required for the screening period will be completed.Ensartinib will be administered at a dose of 200 mg, orally, once daily, for 2 consecutive years. During the first year, efficacy evaluations and safety visits (including physical examinations, laboratory tests, tumor assessments, and quality-of-life assessments) will be conducted every 12 weeks. During the second year and beyond (prior to progression), efficacy evaluations and safety visits will be conducted every 24 weeks.After the study completion by the investigator and the recording of disease progression at each stage, long-term survival follow-up information will be collected every 24 weeks. Patients who discontinue study treatment for reasons other than disease progression (excluding loss to follow-up or death) will continue to undergo objective tumor assessments every 24 weeks to gather information on disease progression. If a patient experiences recurrence within 2 years post-surgery, survival follow-up will be conducted via telephone every 24 weeks after recurrence, continuing until 5 years post-surgery or death.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years;
* ECOG performance status 0-1;
* Postoperative histopathology confirms R0 resection with TNM stage I pulmonary adenocarcinoma;
* Confirmed ALK fusion-positive by FISH, IHC, or NGS;
* No prior systemic treatment after surgery;
* At least one high-risk recurrence factor: poorly differentiated tumor, vascular invasion, wedge resection, visceral pleura involvement, uncertain lymph node status, intrapulmonary dissemination;
* Able to start Ensartinib adjuvant therapy within 4-8 weeks after surgery;
* Hematological, biochemical, and organ function requirements met: Hemoglobin ≥100 g/L; Absolute neutrophil count ≥1.5×10^9/L; Platelet count ≥100×10^9/L; Total bilirubin ≤2 times the upper limit of normal; ALT and AST ≤2.5 times the upper limit of normal; Creatinine ≤1.5 times the upper limit of normal; Creatinine clearance ≥60 mL/min;
* Women of childbearing potential must have a negative urine pregnancy test - within 7 days prior to starting treatment;
* Informed consent obtained from the patient or their legal representative;
* Men and women of childbearing potential must agree to use reliable - contraception from enrollment in the study until 8 weeks after discontinuation of the study drug.

Exclusion Criteria:

* Previous systemic treatment for NSCLC;
* Previous local radiotherapy for NSCLC;
* Unable to take oral medications;
* Known allergy to Ensartinib or any component of this product;
* History of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis requiring steroid treatment, or any clinically evident active interstitial lung disease; baseline CT scan showing idiopathic pulmonary fibrosis;
* Any unstable systemic diseases, including: active infections, uncontrolled hypertension, unstable angina, angina onset within the last 3 months, congestive heart failure (≥ NYHA class II), myocardial infarction (within 6 months prior to enrollment), severe arrhythmias requiring medication, liver, kidney, or metabolic diseases;
* Pregnant or breastfeeding women;
* History of definite neurological or psychiatric disorders, including epilepsy or dementia;
* Any other conditions that the investigator deems unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
2 year disease-free survival rate | up to 2 year
  2-year DFS rate refers to the percentage of patients who remain free of any signs or symptoms of the disease (in this case, cancer) for two years after receiving treatment.

SECONDARY OUTCOMES:
5 year overall survival rate. | up to 5 year
  The 5 year overall survival rate (5-year OS) is a critical measure in clinical oncology, indicating the percentage of patients who are still alive five years after being diagnosed with cancer or starting treatment.
Disease-free survival | up to 5 year
  Disease-free survival (DFS) is a measure used in clinical oncology to describe the length of time after treatment during which a patient remains free from any signs or symptoms of the disease.

IPD SHARING:
Plan to Share IPD: No